CLINICAL TRIAL: NCT01266577
Title: Development of Magnetic Resonance Spectroscopic Imaging Techniques for Imaging Metabolites in Human Brain and Muscle
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 110045; 11-M-0045
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-09-15

CONDITIONS: Brain Mapping; Healthy Volunteer
Keywords: Brain Metabolism; Neurochemistry; Magnetic Resonance Imaging; Mental Illness; Magnetic Resonance Spectroscopy
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One Arm (Other): Subjects receive the same scan
  Interventions: Other: NSR MAGNETOM 7T; Other: 1Tx x 32Rx Head Coil

INTERVENTIONS:
Other: NSR MAGNETOM 7T — The 7 Tesla scanner is a magnet system used to acquire magnetic resonance imaging and spectroscopy
Other: 1Tx x 32Rx Head Coil — Used to perform proton imaging and spectroscopy in the human heads.

SUMMARY:
Background:

- Magnetic resonance imaging (MRI) is a widely used scanning technique to obtain images of the human body and evaluate activity in the brain. A particular MRI method called magnetic resonance spectroscopy (MRS) can be used to study brain chemistry as well, which may help researchers who are studying new treatments for psychiatric illnesses. Researchers are interested in improving current MRI and MRS techniques, as well as developing new MRI and MRS techniques to view and measure brain chemicals and brain activity.

Objectives:

- To implement, develop, and optimize brain chemistry imaging techniques using magnetic resonance imaging and magnetic resonance spectroscopy.

Eligibility:

- Healthy individuals between 18 and 65 years of age.

Design:

* This study will involve a screening visit and a scanning visit at the National Institutes of Health Clinical Center.
* Participants will be screened with a full medical and physical examination, blood and urine tests, and neurological testing.
* During the second visit, participants will have an MRI scan of the brain. (Participants who have received an MRI within the past year will not need to have a second one; the images of the previous scan will be used for this study.) All participants will then have an MRS scan using the same scanning equipment.

DETAILED DESCRIPTION:
Magnetic resonance spectroscopy (MRS) is identical to MRI except that the metabolite signal, rather than the dominant water signal, is measured. Proton (1H) MRS and phosphorous (P) MRS are two powerful spectroscopy methods to measure metabolism in vivo.

By using water suppression techniques, proton MRS can monitor levels of important brain metabolites and neurotransmitters such as N-acetylaspartate (NAA), creatine, choline, lactate, myo-inositol, glutamate, glutamine, gamma aminobutyric acid (GABA), and glutathione.

P MRS can be utilized to measure energy phosphate metabolites of inorganic phosphate (Pi), phosphocreatine (PCr), adenosine diphosphate (ADP), and adenosine triphosphate (ATP) in brain and muscle. In addition, phosphocholine (PC), phosphoethanolamine (PE), glycerophosphocholine (GPC) and glyceophosphoethanolamine (GPE) can also be detected in brain tissues.<TAB>

This protocol proposes three main goals. First, to implement and optimize current proton and P MRS methods published in the literature for the imaging of metabolites in human brain and muscle. Second, to further develop new methods for use in similar brain and muscle MRS applications. Third, to exchange MRS data with other studies in order to provide data analysis and quality control for the studies under this, other NIH, or outside protocols.

To develop and optimize in vivo MRS methods, 300 healthy volunteers will be recruited over a period of ten years. The subjects will be aged 18-65 years, and include representative numbers of males, females, and minorities.

The experiments will be performed on the GE 3T, Siemens 3T and 7T MRI scanners located at the NIH In Vivo NMR Research Center. In the first portion of the study, a clinical MRI will be performed to ensure the subject has no abnormal brain conditions. In the second portion of the study, MRS scans will be performed in various system and pulse parameter combinations. No medications will be involved. Total scan time during the MRS scan will be one to two hours long.

We expect to obtain high quality proton and/or phosphorous spectroscopy imaging from healthy volunteers that will help establish accurate and reliable spectroscopy methods for clinical investigators to perform non-invasive studies of psychiatric, neurological disorders, and other diseases in human brain or muscle.

ELIGIBILITY:
* INCLUSION CRITERIA:
* 18-65 years of age
* able to give written informed consent
* healthy based on medical history and physical exam
* enrolled in Protocol 01-M-0254 or Protocol 17-M-0181

EXCLUSION CRITERIA:

* Any current Axis 1 diagnosis
* Clinically significant laboratory abnormalities
* Positive HIV test
* Metallic foreign bodies that would be affected by the magnetic resonance imaging (MRI) magnet, or fear of enclosed spaces likely to make the subject unable to undergo an MRI scan.
* History of neurological illness or injury with the potential to affect study data interpretation, such as multiple sclerosis, Parkinson s disease, seizure disorder or traumatic brain injury
* Inability to lie flat on camera bed for about two and a half hours
* Pregnant or breastfeeding
* Current substance use disorder based on DSM-5
* NIMH employees and staff and their immediate family members will be excluded from the study per NIMH policy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-01-27 (Actual); Primary Completion 2026-01-24 (Estimated); Study Completion 2026-10-23 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the quality of the MR spectroscopy which includes spectrum signal-to-noise (SNR) ratio, spectral lineshape, linewidth, and resolution. | prospective and ongoing
  to obtain more accurate and reliable MRS data from the human brain and muscle

SECONDARY OUTCOMES:
The secondary outcome is the performance improvements of the scanner hardware, software and methodology. | prospective and ongoing
  to obtain more accurate and reliable MRS data from the human brain and muscle

CONTACTS AND LOCATIONS:
Overall Officials: Li An, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] An L, Shen J. In vivo magnetic resonance spectroscopy by transverse relaxation encoding with narrowband decoupling. Sci Rep. 2023 Jul 27;13(1):12211. doi: 10.1038/s41598-023-39375-0. PMID 37500714
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2011-M-0045.html